CLINICAL TRIAL: NCT06721468
Title: Increasing Trout Consumption in Young Children and Families for Cognitive and Mental Health Benefit
Brief Title: Trout Consumption in Young Children and Families and Brain Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-033
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Change; Well-Being, Psychological
Keywords: Trout; Children; Child-Centered Nutrition Phrases; Cognition; Emotional well-being; Sensory evaluation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Objective 1: Two untrained consumer panels will provide sensory evaluation on three different strains of trout (fish-meal diet, CX line, CLX line).
  Objective 2: A within subjects, pre/post design will be employed to compare the effect of repeated exposure (RE) and repeated exposure plus child centered nutrition phrases (RE+CCNP) on eating behaviors of children 4-6 years of age.
  Objective 3: A 12-week quasi-experimental design will be employed to capture the translational impact of repeated exposure and nutrition education to the home setting on intake of whole CX line trout and the effect on adult and youth cognitive and emotional wellbeing outcomes. A control and three treatment groups will be recruited from a convenience sample of Eat Smart Idaho participants in northern and south central Idaho.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Objective 1: Sensory Evaluation (Experimental): three different strains of trout (fish-meal diet, CX line, CLX line)
  Interventions: Other: Trout
- Objective 2: Repeated Exposure (Experimental): 2 oz of trout each week for 10 weeks
  Interventions: Other: Trout
- Objective 2: Repeated Exposure Plus Child-Centered Nutrition Phrases (Experimental): 2 oz of trout each week plus exposure to positive nutrition message about trout each week for 10 weeks
  Interventions: Other: Trout; Other: Child-centered nutrition phrases
- Objective 2: Puzzle Game (Placebo Comparator): Exposure to a puzzle game each week for 10 weeks
  Interventions: Other: Puzzle
- Objective 3: Eat Smart Idaho (No Intervention): Only receive Eat Smart Idaho's standard 6-lesson in-person series of classes
- Objective 3: Child-Centered Nutrition Phrases (Experimental): Receive Eat Smart Idaho's standard 6-lesson in-person series of classes AND asked to view an online trout-specific nutrition education and recipe preparation video series, "About Trout! Pond to Plate."
  Interventions: Other: Child-centered nutrition phrases
- Objective 3: Repeated Exposure (Experimental): Receive Eat Smart Idaho's standard 6-lesson in-person series of classes AND receive 2 servings of trout per week for 12 weeks, to prepare at home and consume (2 oz. serving for child and 4 oz. serving for adult).
  Interventions: Other: Trout
- Objective 3: Repeated Exposure Plus Child Centered Nutrition Phrases (Experimental): Receive Eat Smart Idaho's standard 6-lesson in-person series of classes, AND receive 2 servings of trout per week for 12 weeks, to prepare at home and consume (2 oz. serving for child and 4 oz. serving for adult), AND asked to view an online trout-specific nutrition education and recipe preparation video series, "About Trout! Pond to Plate."
  Interventions: Other: Trout; Other: Child-centered nutrition phrases

INTERVENTIONS:
Other: Trout — rainbow trout
  Arms: Objective 1: Sensory Evaluation; Objective 2: Repeated Exposure; Objective 2: Repeated Exposure Plus Child-Centered Nutrition Phrases; Objective 3: Repeated Exposure; Objective 3: Repeated Exposure Plus Child Centered Nutrition Phrases
Other: Child-centered nutrition phrases — learn the phrase, "trout helps your brain so you can learn and play" either through researcher introduction or completing the "About Trout! Pond to Plate" curriculum
  Arms: Objective 2: Repeated Exposure Plus Child-Centered Nutrition Phrases; Objective 3: Child-Centered Nutrition Phrases; Objective 3: Repeated Exposure Plus Child Centered Nutrition Phrases
Other: Puzzle — presented with a puzzle to solve each week
  Arms: Objective 2: Puzzle Game

SUMMARY:
Regular fish consumption may support brain health. Trout lines developed in Idaho contain higher levels of omega-3 fatty acids, nutrients important for human cognition and mental wellbeing. Developed to support aquaculture sustainability, consumer preferences and human health benefits of these fish are unknown. The long-term goal of this project is to utilize nutrition education strategies to increase adult and child consumption of fish to improve brain health as measured by cognitive and emotional wellbeing. Research objectives and activities include, (1) adult and child consumer panels to provide sensory evaluation on three strains of trout, (2) effects of repeated exposure (RE) and child-centered nutrition phrases (CCNP) on eating behaviors and brain health will be determined using one control and two treatment groups of children in childcare settings, (3) effects of nutrition education, incorporating CCNP and fish preparation techniques, and RE targeting family meals on eating behaviors of children and brain health of adults and children will be determined using four treatment groups in the home setting.

DETAILED DESCRIPTION:
Regular fish consumption may support brain health. Trout lines developed in Idaho contain higher levels of omega-3 fatty acids, nutrients important for human cognition and mental wellbeing. Developed to support aquaculture sustainability, consumer preferences and human health benefits of these fish are unknown. The long-term goal of this integrated project is to utilize nutrition education strategies to increase adult and child consumption of fish to improve brain health as measured by cognitive and emotional wellbeing. The long-term impact of this project addresses the key knowledge gap in understanding strategies to increase fish consumption in children and adults, which has the positive implication to improve adult and child cognitive and emotional wellbeing. As knowledge of the health benefits of foods such as fish, may not result in increased consumption, this study can provide evidence of repeated exposure and applied educational tools to facilitate consumption by children and adults. Results from this study will fill the gap to provide greater knowledge of cognitive and emotional wellbeing health benefits of fish consumption and strategies for increasing adult and children's fish consumption. A greater intake of fish not only has the potential to contribute to improved population health outcomes, but also has a probable role in sustainability of US agriculture and food systems through promotion of this cost effective source of protein. In addition, better understanding the sensory perceptions of consumers in relation to fish with varied diets is an important step in identifying additional strategies to grow the aquaculture industry. The specific lines of trout being developed at the Hagerman facility do have a focus on sustainability through feeding plant-based diets rather than the traditional fish meal diet, which is less sustainable and more taxing on the aquaculture industry. Having the data on consumer acceptance, and evidence to support nutrition education strategies to increase liking, and consumption of these lines of trout will contribute to the overall sustainability goals.

ELIGIBILITY:
Inclusion Criteria:

* Objective 1: Children 3-6 years of age, adults age 18+, English speaking
* Objective 2: Children 4-6 years of age, English speaking
* Objective 3: Children 4-9 years of age AND parent/guardian, English or Spanish speaking, access to internet, currently eat fish less than twice per week

Exclusion Criteria:

* allergy or dietary restriction preventing consuming fish

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in liking from baseline to 12-weeks | Change from baseline liking at 12-weeks
  subjects rate their liking of trout on a 3-point scale (yummy, just okay, yucky)
Change in intake from baseline to 12-weeks | Change from baseline intake at 12-weeks
  Subjects are offered 2oz of trout each week for 12 weeks. Trout servings are weighed pre/post consumption as a proxy of intake.
Change in cognition composite score from baseline to 12-weeks | Change from baseline cognition composite score at 12-weeks
  Subjects complete a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Early childhood cognition composite score is derived from scores on tthe Dimensional Change Card Sort, Flanker, Picture Sequence Memory, Picture Vocabulary, and Speeded Matching tests.
Change in emotion score from baseline to 12-weeks | Change from baseline emotion score at 12-weeks
  Subjects complete a battery of computerized self-reported or parent proxy questionnaires using the NIHToolbox for Assessment of Neurological and Behavioral Function.
Difference in liking among three trout strains | measured 1 time upon enrollment
  subjects rate their liking of three different trout strains

SECONDARY OUTCOMES:
Change in fluid cognition composite score from baseline to 12-weeks | Change from baseline cognition composite score at 12-weeks
  Subjects complete a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Fluid cognition composite score is derived from scores on the dimensional change card sort, flanker, picture sequence memory, list sorting, and pattern comparison tests.

CONTACTS AND LOCATIONS:
Overall Officials: Annie J Roe, PhD, Principal Investigator — University of Idaho
Locations (2):
- United States (2):
  - University of Idaho, Moscow, Idaho
  - Washington State University, Pullman, Washington

IPD SHARING:
Plan to Share IPD: No
Persons requesting the data will be required to obtain and share IRB approval and to sign a data sharing agreement. Data will be made available one year after the primary manuscripts detailing the major outcomes of the study are published.